CLINICAL TRIAL: NCT01231620
Title: A Phase III International, Randomized, Double-blind, Double-dummy Study to Evaluate the Efficacy and Safety of 300 mg or 600 mg of Intravenous Zanamivir Twice Daily Compared to 75 mg of Oral Oseltamivir Twice Daily in the Treatment of Hospitalized Adults and Adolescents With Influenza
Brief Title: A Study of Intravenous Zanamivir Versus Oral Oseltamivir in Adults and Adolescents Hospitalized With Influenza
Acronym: ZORO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114373
Record Dates: First submitted 2010-10-28; First posted 2010-11-01 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-03

CONDITIONS: Influenza, Human
Keywords: Seasonal Influenza; Pandemic; Orthomyxoviridae Infections; Influenza; Influenza A Virus, H1N1 Subtype; Enzyme Inhibitors; Influenza, seasonal; Respiratory Tract Diseases; Zanamivir; Pharmacologic Actions; Antiviral Agents; Anti-Infective Agents; H1N1; Neuraminidase inhibitor; Influenza B virus
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections; Respiratory Tract Diseases | interventions — Zanamivir; Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intravenous (IV) Zanamivir 300mg Twice Daily (Experimental): 300mg of IV zanamivir infusion twice daily plus oral oseltamivir placebo twice daily
  Interventions: Drug: Zanamivir; Drug: Placebo to match oseltamivir
- Intravenous (IV) Zanamivir 600mg Twice Daily (Experimental): 600mg of IV zanamivir infusion twice daily plus oral oseltamivir placebo twice daily
  Interventions: Drug: Zanamivir; Drug: Placebo to match oseltamivir
- Oral Oseltamivir 75mg Twice Daily (Active Comparator): 75mg oral oseltamivir twice daily plus intravenous placebo zanamivir twice daily
  Interventions: Drug: Placebo to match zanamivir; Drug: Oseltamivir

INTERVENTIONS:
Drug: Zanamivir — Zanamivir aqueous solution, 10 mg/mL, will be provided as a single use, sterile clear, colorless preparation in 20 mL clear glass vials.
  Other Names: Relenza
  Arms: Intravenous (IV) Zanamivir 300mg Twice Daily; Intravenous (IV) Zanamivir 600mg Twice Daily
Drug: Placebo to match zanamivir — Placebo to match IV zanamivir will be provided as a normal saline solution of a matched volume.
  Arms: Oral Oseltamivir 75mg Twice Daily
Drug: Oseltamivir — Oseltamivir will be provided as over-encapsulated 75 mg capsules.
  Other Names: Tamiflu
  Arms: Oral Oseltamivir 75mg Twice Daily
Drug: Placebo to match oseltamivir — Placebo to match oral oseltamivir will be provided as capsules with a common excipient of appropriate quality.
  Arms: Intravenous (IV) Zanamivir 300mg Twice Daily; Intravenous (IV) Zanamivir 600mg Twice Daily

SUMMARY:
The purpose of this study is to test the safety and efficacy of zanamivir given intravenously and how well it works at two different doses in hospitalized adolescents and adults with flu. Zanamivir will be compared with oseltamivir, which is used for treating flu.

DETAILED DESCRIPTION:
The recent influenza pandemic has highlighted the need for alternative formulations for anti-influenza therapies. This will be an international Phase III, double-blind, double-dummy, 3-arm study to evaluate the efficacy, antiviral activity and safety of IV zanamivir 600 mg twice daily compared to oral oseltamivir 75 mg twice daily, and 600 mg IV zanamivir twice daily compared to 300 mg IV zanamivir for 5 days in hospitalized subjects with laboratory confirmed or suspected influenza infection. For a given subject, the initial 5-day treatment course may be extended for up to 5 additional days if clinical symptoms or patient characteristics as assessed by the investigator warrant further treatment. Alternatively, if the investigator considers that a subject is failing to improve clinically on their randomized treatment, the investigator can choose to initiate the switch/rescue option (600 mg IV zanamivir twice daily) on any day from Day 6 through Day 10 for up to an additional 5 days of treatment. On switching treatments, subjects complete a maximum of 14 days of treatment and are followed-up to Post-Treatment +28 Days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 16 years; a female is eligible to enter and participate in the study if she is:

  1. of non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post- menopausal); or,
  2. of child-bearing potential, has a negative pregnancy test at Baseline, and agrees to use protocol specified methods of birth control while on study.
* Vital signs criteria defined as 3 or more of the following at Baseline:

  1. Presence of fever [oral temperature of 38°C or equivalent] at Baseline. However, this requirement is waived if the subject has a history of fever within in the 24 hours prior to Baseline; or, if the subject reported symptoms of feverishness at some time during the 48 hours prior to Baseline.

     AND at least 2 out of the following 4:
  2. Oxygen saturation <95% on room air by trans-cutaneous method or need for any supplemental oxygenation or ventilatory support, or increase in oxygen supplementation requirement of ≥2 litres for subjects with chronic oxygen dependency. For those subjects with a history of chronic hypoxia (without supplemental oxygen), an oxygen saturation of at least 3% below the patient's historical baseline oxygen saturation will satisfy this criterion.
  3. Respiration rate >24 breaths per minute. For those subjects who require ventilatory support or oxygen supplementation, this requirement is waived.
  4. Heart rate >100 beats per minute.
  5. Systolic blood pressure <90 mmHg.
* Onset of influenza symptoms within 6 days prior to study enrolment. Symptoms may include cough, dyspnea, sore throat, feverishness, myalgias, headache, nasal symptoms (rhinorrhea, congestion), fatigue, diarrhea, anorexia, nausea and vomiting.
* Clinical symptoms of influenza with positive influenza diagnostic test result or strong suspicion of influenza illness based on clinical symptoms and local surveillance information.
* Subjects willing and able to give written informed consent to participate in the study and to adhere to the procedures stated in the protocol, or legally acceptable representative willing and able to give written informed consent on behalf of the subject for minors, unconscious adults and those incapable of consenting themselves due to their medical condition, or included as permitted by local regulatory authorities, IRB/IECs or local laws.
* Severity of any medical illness that, in the Investigator's judgement, justifies hospitalization of the subject for treatment and supportive care
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category

Exclusion Criteria:

* Subjects who have taken more than a total of 3 days (6 doses) of approved anti-influenza therapy in the period from onset of symptoms and prior to enrolment.
* Subjects who, in the opinion of the investigator, are not likely to survive beyond 48 hours from Baseline.
* Subjects who are considered to require concurrent therapy with another influenza antiviral medication.
* Subjects who are known or suspected to be hypersensitive to any component of the study medications.
* Subjects with creatinine clearance ≤10 mL/min who are not being treated with continuous renal replacement therapy (CRRT).
* Subjects who require Extra Corporeal Membrane Oxygenation (ECMO) at Baseline
* Subjects who require routine/intermittent hemodialysis or continuous peritoneal dialysis (due to inability to provide appropriate dosing schedule for oseltamivir) at Baseline. CRRT modalities are allowed.
* Liver toxicity criteria based on local laboratory results obtained within 24 hours of Baseline:

  1. ALT or AST 3xULN and bilirubin 2xULN
  2. ALT 5xULN
* Underlying chronic liver disease with evidence of severe liver impairment.
* History of severe cardiac disease or clinically significant arrhythmia (either on ECG or by history) which, in the opinion of the Investigator, will interfere with the safety of the individual subject.
* Females who are pregnant or are breastfeeding.
* Treatment with investigational parenteral anti-influenza drugs (IV peramivir, IV zanamivir or IV oseltamivir) in the 4 weeks prior to Baseline.
* French and Korean subjects: the French or Korean subject has participated in any study using an investigational drug during the previous 30 days.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Start 2011-01-15 (Actual); Primary Completion 2015-03-18 (Actual); Study Completion 2015-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (154):
- United States (40):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Escondido, California
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, La Mesa, California
  - GSK Investigational Site, Oceanside, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Stamford, Connecticut
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Sunrise, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Idaho Falls, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Oak Park, Illinois
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Council Bluffs, Iowa
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Royal Oak, Michigan
  - GSK Investigational Site, Troy, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Valhalla, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Bismarck, North Dakota
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Bethlehem, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Roanoke, Virginia
  - GSK Investigational Site, Marshfield, Wisconsin
- Australia (8):
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Bedford Park, South Australia
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Perth, Western Australia
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
- Brazil (2):
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, São Paulo
- Canada (7):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Chicoutimi, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- China (13):
  - GSK Investigational Site, Haikou, Hainan
  - GSK Investigational Site, Changsha, Hunan
  - GSK Investigational Site, Nanchang, Jiangxi
  - GSK Investigational Site, Changchun, Jilin
  - GSK Investigational Site, Xi'an, Shaanxi
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin
- GSK Investigational Site, Bogotá, Colombia
- Czechia (4):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Brno-Bohunice
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Prague
- Denmark (3):
  - GSK Investigational Site, Aarhus N
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, Odense C
- France (6):
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Nîmes
  - GSK Investigational Site, Orléans
  - GSK Investigational Site, Poitiers
  - GSK Investigational Site, Tours
- Germany (5):
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Homburg, Saarland
- Greece (2):
  - GSK Investigational Site, Chaïdári
  - GSK Investigational Site, Goudi, Athens
- Hong Kong (3):
  - GSK Investigational Site, Kwun Tong
  - GSK Investigational Site, Shatin
  - GSK Investigational Site, Tuenmen
- Hungary (5):
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Kaposvár
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Székesfehérvár
  - GSK Investigational Site, Szombathely
- India (5):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Civil Lines
  - GSK Investigational Site, Lucknow
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Trivandrum
- Mexico (5):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, San Nicolás de los Garza, Nuevo León
  - GSK Investigational Site, Cuautitlán, Estado de México, State of Mexico
  - GSK Investigational Site, Aguascalientes
  - GSK Investigational Site, Chihuahua City
- GSK Investigational Site, Nijmegen, Netherlands
- New Zealand (5):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, Hastings
  - GSK Investigational Site, Newtown
- Norway (2):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Trondheim
- Poland (4):
  - GSK Investigational Site, Chorzów
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Trzebnica
  - GSK Investigational Site, Warsaw
- Russia (3):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Smolensk
- Slovakia (2):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Martin
- South Africa (6):
  - GSK Investigational Site, Middelburg, Mpumalanga
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Die Wilgers
  - GSK Investigational Site, Les Marais
  - GSK Investigational Site, Panorama
  - GSK Investigational Site, Worcester
- South Korea (4):
  - GSK Investigational Site, Guro Gu
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Kangwon-do
  - GSK Investigational Site, Seoul
- Spain (9):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Granada
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Pama de Mallorca
- GSK Investigational Site, Taipei, Taiwan
- GSK Investigational Site, Bangkok, Thailand
- United Kingdom (4):
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Cardiff
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] van Duijnhoven W, Van Dromme I, Haesendonckx S, Witek J, Leopold L. The Hospital Recovery Scale: A clinically useful endpoint in patients hospitalized with influenza. Contemp Clin Trials. 2022 Dec;123:106952. doi: 10.1016/j.cct.2022.106952. Epub 2022 Oct 3. PMID 36202198
- [Derived] Marty FM, Vidal-Puigserver J, Clark C, Gupta SK, Merino E, Garot D, Chapman MJ, Jacobs F, Rodriguez-Noriega E, Husa P, Shortino D, Watson HA, Yates PJ, Peppercorn AF. Intravenous zanamivir or oral oseltamivir for hospitalised patients with influenza: an international, randomised, double-blind, double-dummy, phase 3 trial. Lancet Respir Med. 2017 Feb;5(2):135-146. doi: 10.1016/S2213-2600(16)30435-0. Epub 2017 Jan 14. PMID 28094141
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 114373 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114373 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114373 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114373 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114373 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114373 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114373 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Male and female adult and adolescent participants >=16 years of age hospitalized with documented influenza or suspected influenza were eligible for enrollment. A total of 626 participants were randomized, and 615 participants were included in the Intent-to-Treat Exposed (ITT-E) Population (pop)
Groups:
- IV Zanamivir 300 mg: Participants >=16 years of age received intravenous (IV) zanamivir 300 milligrams (mg) twice daily, adjusted for renal function for 5-10 days.
- IV Zanamivir 600 mg: Participants >=16 years of age received IV zanamivir 600 mg twice daily, adjusted for renal function for 5-10 days
- Oral Oseltamivir 75 mg: Participants >=16 years of age received oral oseltamvir 75 mg twice daily, adjusted for renal function for 5-10 days.
Period: Overall Study
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Started | 201 | 209 | 205
Completed | 175 | 178 | 166
Not Completed | 26 | 31 | 39
Not completed — Physician Decision | 3 | 5 | 10
Not completed — Death | 12 | 14 | 11
Not completed — Adverse Event | 2 | 2 | 1
Not completed — Withdrawal by Subject | 6 | 6 | 8
Not completed — Lost to Follow-up | 3 | 4 | 9

BASELINE CHARACTERISTICS:
Groups:
- IV Zanamivir 300 mg: Participants >=16 years of age received IV zanamivir 300 mg twice daily, adjusted for renal function for 5-10 days.
- Total: Total of all reporting groups
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg | Total
Number analyzed (Participants) | 201 | 209 | 205 | 615
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.2 (18.88) | 57.3 (17.39) | 55.9 (18.7) | 56.2 (18.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 86 | 117 | 285
  Male | 119 | 123 | 88 | 330
Race/Ethnicity, Customized [Number; unit: Participants]
  African American or African Heritage | 12 | 4 | 10 | 26
  American Indian or Alaskan Native | 3 | 2 | 4 | 9
  Asian - Central South Asian | 10 | 15 | 13 | 38
  Asian - East Asian Heritage | 12 | 18 | 13 | 43
  Asian - South East Asian Heritage | 6 | 4 | 7 | 17
  Native Hawaiian or Other Pacific | 2 | 1 | 0 | 3
  White - Arabic or North African | 4 | 3 | 3 | 10
  White -White or Caucasian or European | 150 | 162 | 154 | 466
  Unknown | 1 | 0 | 1 | 2
  Mixed Race | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Clinical Response (TTCR) in Participants With Confirmed Influenza
Description: Clinical response is defined as the resolution of at least 4 of the 5 vital signs (temperature, oxygen saturation, respiratory status, heart rate, systolic blood pressure) within the respective resolution criteria, maintained for at least 24 hours, or hospital discharge, whichever occurred first. This analysis was performed for Influenza positive population, for those with symptom onset less than or equal to (<=) 4 days, and for those on mechanical (mech) ventilation or in intensive care unit (ICU). 99 days is censored time for the participants who did not achieve TTCR.
Time Frame: Up to 42 days
Population: ITT-E population comprised of all randomized participants who received at least one dose of investigational product. The Influenza positive population (IPP) is comprised of all participants in the ITT-E population with proven influenza infection.
Measure: Median (Full Range); unit: Days
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 163 | 162 | 163
Days | 5.87 [0.12 to 99.90] | 5.14 [0.23 to 99.90] | 5.63 [0.03 to 99.90]
Statistical Analysis 1: Comparison: IV Zanamivir 300 mg vs IV Zanamivir 600 mg; Test type: Superiority or Other; p = 0.25, Wilcoxon rank sum; Median Difference (Final Values) = -0.73, 95% CI 2-sided [-1.79 to 0.75] — IV Zanamivir 300 mg versus IV Zanamivir 600 mg
Statistical Analysis 2: Comparison: IV Zanamivir 600 mg vs Oral Oseltamivir 75 mg; Test type: Superiority or Other; p = 0.39, Wilcoxon rank sum; Median Difference (Final Values) = -0.48, 95% CI 2-sided [-2.11 to 0.97] — Oral oseltamivir 75 mg versus IV Zanamivir 600 mg

2. Secondary Outcome: Percentage of Participants With Respiratory Improvement
Description: Respiratory Status (RS) is a component of TTCR. Response criteria included the return to the pre-morbid oxygen requirement (participants with chronic oxygen use), a need for supplemental oxygen (administered by any modality: ventilator, non-invasive ventilation, facemask, facetent, nasal canula, etc.) to no need for supplemental oxygen, or a respiratory rate of =<24 breaths/minute (without supplemental oxygen). Data are presented as the percentage of participants achieving respiratory improvement.
Time Frame: Up to 42 days
Population: IPP Population
Measure: Number; unit: Percentage of participants
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 163 | 162 | 163
Percentage of participants | 77 | 78 | 74
Statistical Analysis 1: Comparison: IV Zanamivir 300 mg vs IV Zanamivir 600 mg; Test type: Superiority or Other; p = 0.506, Wei-Johnson method
Statistical Analysis 2: Comparison: IV Zanamivir 600 mg vs Oral Oseltamivir 75 mg; Test type: Superiority or Other; p = 0.41, Wei-Johnson method

3. Secondary Outcome: Number of Participants With All Cause and Attributable Mortality at Day 14, at Day 28, and at the End of Study Visit
Description: The number of participants who died on or before Day 14, Day 28, and the End of Study Visit were summarized.
Time Frame: On or before Day 14, Day 28, End of Study Visit (assessed up to 42 days)
Population: IPP Population
Measure: Count of Participants; unit: Participants
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 163 | 162 | 163
Participants
  Died on or before Study Day 14: all cause | 5 | 8 | 5
  Died on or before Study Day 28: all cause | 8 | 9 | 9
  Died while on-study: all cause | 10 | 12 | 10
  Died on or before Study Day 14: attributable | 3 | 4 | 4
  Died on or before Study Day 28: attributable | 5 | 5 | 5
  Died while on-study: attributable | 5 | 6 | 6

4. Secondary Outcome: Change From Baseline in the Katz Activities of Daily Living (ADL) Score and Each ADL Activity Score
Description: The Katz ADL scores were collected for bathing, dressing, toileting, transferring, continence, and feeding activities and were assessed once daily during the treatment period/hospitalization and once at each post-treatment Clinic Visit. For the six individual activities, a score of 1 indicates independence, and a score of 0 indicates dependence. The total score is generated by adding the scores of all six activities. A total score of 6 indicates that the participant was independent; a total score of 0 indicates that the participant was very dependent. Baseline is defined as the pre-dose value collected on Study Day 1. Change from Baseline is defined as the difference at each time point (Day 5/6, and Day 10/11, and last day S/R if treatment was extended beyond 5 days) and the end of the study (post-treatment [PT] +28 Days) compared to Baseline.
Time Frame: Baseline (Day 1) and up to 42 days
Population: IPP population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on the scale
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 163 | 162 | 163
Scores on the scale
  Total Score Day 5/6: number analyzed (Participants) | 149 | 150 | 139
  Total Score Day 5/6 | 1.07 (1.959) | 0.93 (1.782) | 0.78 (1.837)
  Total Score Day 10/11: number analyzed (Participants) | 16 | 6 | 12
  Total Score Day 10/11 | 0.88 (1.746) | 0.5 (0.837) | -0.08 (3.029)
  Total Score Last Day of S/R: number analyzed (Participants) | 5 | 2 | 8
  Total Score Last Day of S/R | 0.2 (2.49) | -3.0 (4.243) | 0.75 (1.165)
  Total Score PT+28 Day: number analyzed (Participants) | 138 | 134 | 120
  Total Score PT+28 Day | 2.13 (2.234) | 1.72 (2.342) | 1.98 (2.142)
  Bathing: DAY 5/6: number analyzed (Participants) | 149 | 150 | 139
  Bathing: DAY 5/6 | 0.24 (0.488) | 0.19 (0.429) | 0.18 (0.438)
  Bathing: DAY 10/11: number analyzed (Participants) | 16 | 6 | 12
  Bathing: DAY 10/11 | 0.19 (0.403) | 0.0 (0.0) | 0.0 (0.426)
  Bathing: Last Day of S/R: number analyzed (Participants) | 5 | 2 | 8
  Bathing: Last Day of S/R | 0.2 (0.447) | -0.5 (0.707) | 0.0 (0.0)
  Bathing: PT + 28 DAYS: number analyzed (Participants) | 138 | 134 | 120
  Bathing: PT + 28 DAYS | 0.43 (0.498) | 0.34 (0.505) | 0.39 (0.507)
  Dressing DAY 5/6: number analyzed (Participants) | 149 | 150 | 139
  Dressing DAY 5/6 | 0.23 (0.481) | 0.21 (0.438) | 0.14 (0.427)
  Dressing: Day 10/11: number analyzed (Participants) | 16 | 6 | 12
  Dressing: Day 10/11 | 0.13 (0.342) | 0.0 (0.0) | -0.08 (0.515)
  Dressing: Last Day of S/R: number analyzed (Participants) | 5 | 2 | 8
  Dressing: Last Day of S/R | 0.2 (0.447) | -0.5 (0.707) | 0.13 (0.354)
  Dressing:PT+28 Day: number analyzed (Participants) | 138 | 134 | 120
  Dressing:PT+28 Day | 0.42 (0.495) | 0.37 (0.515) | 0.41 (0.494)
  Toileting: DAY 5/6: number analyzed (Participants) | 149 | 150 | 139
  Toileting: DAY 5/6 | 0.19 (0.456) | 0.19 (0.439) | 0.14 (0.409)
  Toileting: Day 10/11: number analyzed (Participants) | 16 | 6 | 12
  Toileting: Day 10/11 | 0.13 (0.342) | 0.33 (0.516) | 0.08 (0.515)
  Toileting: Last Day of S/R: number analyzed (Participants) | 5 | 2 | 8
  Toileting: Last Day of S/R | 0.2 (0.447) | -0.5 (0.707) | 0.0 (0.535)
  Toileting: PT+28 Day: number analyzed (Participants) | 138 | 134 | 120
  Toileting: PT+28 Day | 0.4 (0.491) | 0.32 (0.514) | 0.37 (0.484)
  Transferring: DAY 5/6: number analyzed (Participants) | 149 | 150 | 139
  Transferring: DAY 5/6 | 0.28 (0.505) | 0.23 (0.451) | 0.17 (0.41)
  Transferring: Day 10/11: number analyzed (Participants) | 16 | 6 | 12
  Transferring: Day 10/11 | 0.19 (0.403) | 0.17 (0.408) | 0.08 (0.515)
  Transferring: Last Day of S/R: number analyzed (Participants) | 5 | 2 | 8
  Transferring: Last Day of S/R | 0.0 (0.707) | -0.5 (0.707) | 0.25 (0.463)
  Transferring: PT+28 Day: number analyzed (Participants) | 138 | 134 | 120
  Transferring: PT+28 Day | 0.45 (0.499) | 0.36 (0.526) | 0.4 (0.492)
  Continence: DAY 5/6: number analyzed (Participants) | 149 | 150 | 139
  Continence: DAY 5/6 | 0.07 (0.322) | 0.05 (0.314) | 0.07 (0.374)
  Continence: Day 10/11: number analyzed (Participants) | 16 | 6 | 12
  Continence: Day 10/11 | 0.13 (0.342) | 0.0 (0.0) | -0.08 (0.669)
  Continence: Last Day of S/R: number analyzed (Participants) | 5 | 2 | 8
  Continence: Last Day of S/R | -0.2 (0.447) | -0.5 (0.707) | 0.13 (0.354)
  Continence: PT+28 Day: number analyzed (Participants) | 138 | 134 | 120
  Continence: PT+28 Day | 0.22 (0.431) | 0.16 (0.422) | 0.23 (0.439)
  Feeding: Day 5/6: number analyzed (Participants) | 149 | 150 | 139
  Feeding: Day 5/6 | 0.07 (0.331) | 0.07 (0.309) | 0.08 (0.382)
  Feeding: Day 10/11: number analyzed (Participants) | 16 | 6 | 12
  Feeding: Day 10/11 | 0.13 (0.342) | 0.0 (0.0) | -0.08 (0.669)
  Feeding: Last Day of S/R: number analyzed (Participants) | 5 | 2 | 8
  Feeding: Last Day of S/R | -0.2 (0.447) | -0.5 (0.707) | 0.25 (0.463)
  Feeding: PT+28 Day: number analyzed (Participants) | 138 | 134 | 120
  Feeding: PT+28 Day | 0.21 (0.409) | 0.17 (0.416) | 0.19 (0.395)

5. Secondary Outcome: Median Time to Return to Pre-morbid Functional Status as Measured by the Katz ADL Score and Each ADL Activity Score
Description: Pre-morbid functional status is defined as the best functional status in the 4 weeks prior to enrolment. Median time to return to pre-morbid functional status was assessed via the Katz ADL score (bathing, dressing, toileting, transferring, continence, and feeding activities). For the six individual activities, a score of 1 indicates independence, and a score of 0 indicates dependence. The total score is generated by adding the scores of all six activities. A total score of 6 indicates that the participant was independent; a total score of 0 indicates that the participant was very dependent.
Time Frame: Up to 42 days
Population: IPP population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Days
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 163 | 162 | 163
Days
  Total score | 2 [2 to 38] | 2 [2 to 37] | 2.5 [2 to 57]
  Bathing | 2 [2 to 38] | 2 [2 to 37] | 2 [2 to 57]
  Dressing | 2 [2 to 38] | 2 [2 to 40] | 2 [2 to 57]
  Toileting | 2 [2 to 38] | 2 [2 to 31] | 2 [2 to 40]
  Transferring | 2 [2 to 38] | 2 [2 to 31] | 2 [2 to 40]
  Continence | 2 [2 to 35] | 2 [2 to 33] | 2 [2 to 31]
  Feeding | 2 [2 to 29] | 2 [2 to 32] | 2 [2 to 36]

6. Secondary Outcome: Number of Participants Who Returned to Their Pre-morbid Functional Status as Assessed Per the Katz ADL Score and Each ADL Activity Score at the End of the Study
Description: Pre-morbid functional status is defined as the best functional status in the 4 weeks prior to enrolment. The number of participants who returned to their pre-morbid functional status at the end of the study assessed per the Katz ADL score (bathing, dressing, toileting, transferring, continence and feeding activities) is summarized.
Time Frame: Up to 42 days
Population: IPP Population
Measure: Count of Participants; unit: Participants
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 163 | 162 | 163
Participants
  Total | 139 | 138 | 130
  Bathing | 135 | 133 | 126
  Dressing | 138 | 135 | 126
  Toileting | 139 | 136 | 130
  Transferring | 140 | 140 | 133
  Continence | 142 | 143 | 139
  Feeding | 145 | 148 | 144

7. Secondary Outcome: Median Time to Return to the Pre-morbid Level of Activity as Measured by the 3-point Scale
Description: Median time to return to pre-morbid level of activity was assessed once daily during treatment/hospitalization and once at each post-treatment assessment and was measured using the 3- point scale (bed rest, limited ambulation, or unrestricted).
Time Frame: Up to 42 days
Population: IPP Population. Participants succeeded in pre-morbid functional status were analyzed.
Measure: Median (Full Range); unit: Days
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 138 | 137 | 135
Days | 5 [2 to 34] | 4 [2 to 31] | 4 [1 to 57]

8. Secondary Outcome: Number of Participants With the Indicated Clinical Symptoms of Influenza
Description: Influenza clinical symptoms included nasal symptoms (rhinorrhea, congestion), feverishness, cough, myalgias, fatigue, diarrhea, anorexia, dyspnea, headache, sore throat, nausea, and vomiting. Influenza symptoms were assessed once daily during inpatient hospitalization and once at each post-treatment assessment.
Time Frame: Up to 42 days
Population: IPP Population
Measure: Count of Participants; unit: Participants
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 163 | 162 | 163
Participants
  Anorexia | 102 | 112 | 123
  Cough | 151 | 150 | 157
  Diarrhea | 64 | 57 | 66
  Dyspnea | 143 | 145 | 152
  Fatigue | 144 | 144 | 148
  Feverishness | 138 | 145 | 136
  Headache | 104 | 102 | 103
  Myalgias | 115 | 117 | 114
  Nasal symptoms (rhinorrhea, congestion) | 118 | 123 | 122
  Nausea | 57 | 51 | 77
  Sore throat | 94 | 115 | 97
  Vomiting | 27 | 23 | 45

9. Secondary Outcome: Median Time of Duration of Clinical Symptoms of Influenza
Description: Influenza clinical symptoms included nasal symptoms (rhinorrhea, congestion), feverishness, cough, myalgias, fatigue, diarrhea, anorexia, dyspnea, headache, sore throat, nausea, and vomiting. Influenza symptoms were assessed once daily during inpatient/hospitalization and once at each post-treatment assessment.
Time Frame: Up to 42 days
Population: IPP Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Days
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 163 | 162 | 163
Days
  Anorexia: number analyzed (Participants) | 102 | 112 | 123
  Anorexia | 5 [1 to 39] | 3 [1 to 46] | 5 [1 to 55]
  Cough: number analyzed (Participants) | 151 | 150 | 157
  Cough | 14 [1 to 39] | 13 [1 to 46] | 15 [1 to 56]
  Diarrhea: number analyzed (Participants) | 64 | 57 | 66
  Diarrhea | 3 [1 to 29] | 2 [1 to 28] | 3 [1 to 23]
  Dyspnea: number analyzed (Participants) | 143 | 145 | 152
  Dyspnea | 7 [1 to 40] | 6 [1 to 43] | 8 [1 to 56]
  Fatigue: number analyzed (Participants) | 144 | 144 | 148
  Fatigue | 11 [1 to 41] | 11 [1 to 44] | 12 [1 to 56]
  Feverishness: number analyzed (Participants) | 138 | 145 | 136
  Feverishness | 2 [1 to 28] | 2 [1 to 29] | 2.5 [1 to 56]
  Headache: number analyzed (Participants) | 104 | 102 | 103
  Headache | 3 [1 to 33] | 3 [1 to 33] | 4 [1 to 56]
  Myalgias: number analyzed (Participants) | 115 | 117 | 114
  Myalgias | 4 [1 to 39] | 3 [1 to 34] | 4 [1 to 56]
  Nasal symptoms: number analyzed (Participants) | 118 | 123 | 122
  Nasal symptoms | 6 [1 to 34] | 4 [1 to 43] | 5.5 [1 to 35]
  Nausea: number analyzed (Participants) | 57 | 51 | 77
  Nausea | 3 [1 to 34] | 2 [1 to 24] | 2 [1 to 28]
  Sore throat: number analyzed (Participants) | 94 | 115 | 97
  Sore throat | 3 [1 to 28] | 2 [1 to 36] | 3 [1 to 35]
  Vomiting: number analyzed (Participants) | 27 | 23 | 45
  Vomiting | 2 [1 to 19] | 1 [1 to 11] | 1 [1 to 20]

10. Secondary Outcome: Number of Participants With Complications of Influenza and Associated Antibiotic Use
Description: The number of participants with complications of influenza and associated antibiotic use were summarized
Time Frame: Up to 42 days
Population: IPP Population
Measure: Count of Participants; unit: Participants
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 163 | 162 | 163
Participants
  Associated use of any antibiotic | 22 | 16 | 29
  Any complication of influenza | 34 | 33 | 41

11. Secondary Outcome: Number of Participants With the Indicated Ventilation Status: Modality of Invasive and Non-invasive Ventilator Support and Oxygen Supplementation
Description: Ventilation status was assessed three times daily during the treatment period/hospitalization. Ventilation status was assessed once daily during inpatient/hospitization and once at each post-treatment clinic visit. The number of participants reported for machine-assisted: extracorporeal membrane oxygenation (ECMO), endotracheal mechanical ventilation, and supplemental oxygen delivery (SOD), no supplemental oxygen (O2) or ventilation support, Respiratory support at "any time (AT) on study" and at Baseline (Day 1) are summarized. Data for the "any time (AT) on study" time point was reported.
Time Frame: Up to 42 days
Population: IPP Population
Measure: Count of Participants; unit: Participants
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 163 | 162 | 163
Participants
  Day 1, Machine-Assisted: ECMO | 0 | 0 | 0
  Day 1, Machine-Assisted: Endotracheal | 28 | 25 | 27
  Day 1, SOD | 96 | 103 | 87
  Day 1, No supplemental O2 or ventilation support | 32 | 29 | 37
  Day 1, Respiratory Support | 34 | 29 | 39
  AT on Study, Machine-Assisted: ECMO | 2 | 0 | 1
  AT on Study, Machine-Assisted: Endotracheal | 36 | 31 | 37
  AT on Study, SOD | 137 | 137 | 128
  AT on Study, No supplemental O2 or ventilation sup | 138 | 135 | 131
  AT on Study, Respiratory Support | 46 | 37 | 50

12. Secondary Outcome: Median Time of Duration of Invasive and Non-invasive Ventilator Support and Oxygen Supplementation
Description: Ventilation status was assessed three times daily during the treatment period/hospitalization. Ventilation status was assessed once daily during inpatient/hospitalization and once at each post-treatment clinic visit.
Time Frame: Baseline (Day 1) and up to 42 days
Population: IPP Population. Only those participants available with the indicated ventilator support or oxygen supplementation were analyzed.
Measure: Median (Full Range); unit: Days
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 163 | 162 | 163
Days
  Ventilator Support: number analyzed (Participants) | 46 | 37 | 50
  Ventilator Support | 9 [0 to 38] | 5.2 [0 to 36] | 8.2 [0 to 36]
  Oxygen Supplementation: number analyzed (Participants) | 137 | 137 | 128
  Oxygen Supplementation | 4.4 [0 to 38] | 4.2 [0 to 43] | 3.7 [0 to 36]

13. Secondary Outcome: Median Time of Duration of Hospitalization and Intensive Care Unit (ICU) Stay
Description: Hospital duration and ICU duration was assessed from the first day of dosing. Hospital duration was calculated as the discharge date minus the admission date + 1. Hospital duration while on study was the earlier of discharge, completion, or withdrawal minus the later of the admission date or the study start date + 1. ICU duration-Modified was calculated as the original ICU duration minus ICU days prior to Study Day 1.
Time Frame: Day 1 to the end of the study (assessed up to 42 days)
Population: IPP population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Days
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 163 | 162 | 163
Days
  Hospitalization | 10 [1 to 108] | 8 [2 to 64] | 9 [1 to 58]
  Hospitalization while on study | 8 [1 to 39] | 6 [1 to 43] | 7 [1 to 39]
  Hospitalization-ICU: number analyzed (Participants) | 72 | 56 | 71
  Hospitalization-ICU | 8 [1 to 41] | 7.5 [1 to 36] | 8 [1 to 36]
  ICU Duration Modified: number analyzed (Participants) | 70 | 54 | 69
  ICU Duration Modified | 7 [1 to 39] | 6 [1 to 36] | 7 [1 to 36]

14. Secondary Outcome: Median Time to the Absence of Fever and Improved Respiratory Status, Oxygen Saturation, Heart Rate, and Systolic Blood Pressure
Description: The absence of fever is defined as a non-axillary temperature recording <=36.6 degrees Celsius axillary, <= 37.2 degrees Celsius oral or <= 37.7 degrees Celsius core. Respiratory Status (RS) response criteria included the return to the pre-morbid oxygen requirement (participants with chronic oxygen use), or the need for supplemental oxygen (administered by any modality: ventilator, non-invasive ventilation, facemask, facetent, nasal canula, etc.) to no need for supplemental oxygen, or a respiratory rate =<24 breaths/minute (without supplemental oxygen). Oxygen saturation response criteria: >=95% (without supplemental oxygen). Heart rate response criteria: =<100 beats/minute. Systolic blood pressure response criteria: >=90 millimeters of mercury. Vital signs were assessed three times daily during the treatment period/hospitalization. Vital signs were assessed once daily during inpatient/hospitization and once at each post-treatment clinic visit.
Time Frame: Baseline (Day 1) and up to 42 days
Population: IPP Population
Measure: Median (Full Range); unit: Days
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 163 | 162 | 163
Days
  Fever | 1.6 [0 to 34] | 0.8 [0 to 14] | 1.5 [0 to 31]
  Oxygen Saturation: number analyzed (Participants) | 98 | 108 | 99
  Oxygen Saturation | 5.3 [0 to 30] | 5.6 [0 to 32] | 4.5 [0 to 25]
  Respiratory status: number analyzed (Participants) | 126 | 126 | 121
  Respiratory status | 3.5 [0 to 31] | 3.6 [0 to 32] | 2.8 [0 to 21]
  Heart rate: number analyzed (Participants) | 156 | 148 | 155
  Heart rate | 0.4 [0 to 28] | 0.4 [0 to 21] | 0.5 [0 to 24]
  Systolic blood pressure: number analyzed (Participants) | 156 | 156 | 154
  Systolic blood pressure | 0.3 [0 to 23] | 0.3 [0 to 14] | 0.3 [0 to 16]

15. Secondary Outcome: Median Time to Virologic Improvement
Description: Virologic improvement is defined as a 2 log drop in viral load or sustained undetectable viral ribonucleic acid (RNA) (on two successive occasions) as measured by quantitative reverse transcriptase-polymerase chain reaction (RT-PCR) from nasopharyngeal samples. Nasopharyngeal swabs were collected daily from Baseline through Day 5. If randomized treatment was continued beyond Day 5, samples were taken on Treatment Days 6, 8, 10 and on the last day of randomized treatment. For participants who utilized the Switch (S)/Rescue (R) option, samples were taken on S/R Day 1, S/R Day 3, S/R Day 5, or S/R Day 6, whichever was the last day of S/R treatment. Nasopharyngeal swabs were taken if the participant was symptomatic and continued to be hospitalized on the Post-Treatment +2, +5, +9, +16, and +28 day assessment.
Time Frame: Baseline (Day 1) and up to 42 days
Population: IPP Population. Only those participants available at the specified time points were analyzed. Data presented is for participants positive at Baseline.
Measure: Median (Full Range); unit: Days
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 163 | 162 | 163
Days
  Influenza A and B: number analyzed (Participants) | 116 | 122 | 129
  Influenza A and B | 3 [2 to 34] | 3 [2 to 35] | 3 [2 to 34]
  Influenza A/H1N1: number analyzed (Participants) | 47 | 42 | 48
  Influenza A/H1N1 | 3 [2 to 13] | 3 [2 to 34] | 3 [2 to 34]
  Influenza A/H3N2: number analyzed (Participants) | 55 | 58 | 61
  Influenza A/H3N2 | 3 [2 to 8] | 3 [2 to 35] | 3 [2 to 11]
  Influenza B: number analyzed (Participants) | 15 | 20 | 21
  Influenza B | 5 [2 to 34] | 3 [2 to 21] | 3 [2 to 12]

16. Secondary Outcome: Change From Baseline in Quantitative Virus Culture From Nasopharyngeal Swabs Positive at Baseline
Description: Nasopharyngeal swabs were collected daily from Baseline through Day 5. If randomized treatment was continued beyond Day 5, samples were taken on Treatment Day 6, Day 8, Day 10, Day 11, and the last day of randomized treatment. For participants who utilized the S/R option, samples were taken on S/R Day1, S/R Day3, S/R Day5, or S/R Day6, whichever was the last day of S/R treatment. Samples were taken if the participant was symptomatic and continued to be hospitalized on the Post-Treatment +2, +5, +9, +16 and +28Day assessment. Viral load was measured by Quantitative Virus Culture, log10 50% Tissue Culture Infectious Dose (TCID50)/milliliter (mL). Baseline is defined as the pre-dose value collected on Study Day 1. Change from Baseline was calculated as the post-Baseline value minus Baseline value .
Time Frame: Baseline (Day 1), Day 3, Day 5, Day 8, Day 10, Day 11 and/or last day of randomized treatment, if randomized treatment was extended beyond 5 days, and S/R Day 5/6 (up to Day 14) if applicable
Population: IPP Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: log10 TCID50/mL
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 163 | 162 | 163
log10 TCID50/mL
  Day 3: number analyzed (Participants) | 78 | 76 | 89
  Day 3 | -2.01 [-5.0 to 0.8] | -2.01 [-4.8 to 1.3] | -2.01 [-5.3 to 2.8]
  Day 5: number analyzed (Participants) | 66 | 69 | 80
  Day 5 | -2.51 [-5.5 to 0.0] | -2.26 [-5.3 to 0.0] | -2.26 [-5.3 to 2.0]
  Day 8: number analyzed (Participants) | 6 | 7 | 10
  Day 8 | -1.64 [-5.5 to 0.0] | -2.01 [-4.3 to -0.3] | -2.26 [-4.3 to 0.0]
  Day 10: number analyzed (Participants) | 4 | 3 | 4
  Day 10 | -3.76 [-5.5 to -0.3] | -0.3 [-1.3 to -0.3] | -2.26 [-3.8 to -1.3]
  Day 11: number analyzed (Participants) | 3 | 3 | 4
  Day 11 | -3.01 [-5.5 to -0.3] | -0.3 [-0.3 to -0.3] | -2.26 [-3.8 to -1.3]
  S/R Day 5: number analyzed (Participants) | 0 | 1 | 1
  S/R Day 5 |  | -4.3 [-4.3 to -4.3] | -3.0 [-3.0 to -3.0]
  S/R Day 6: number analyzed (Participants) | 1 | 1 | 1
  S/R Day 6 | -2.5 [-2.5 to -2.5] | -4.3 [-4.3 to -4.3] | 0.0 [0.0 to 0.0]

17. Secondary Outcome: Change From Baseline Viral Load (Influenza A or B) by qPCR From Nasopharyngeal Swabs Positive at Baseline
Description: Nasopharyngeal swabs were collected daily from Baseline through Day 5. If randomized treatment was continued beyond Day 5, samples were taken on Treatment Day 6, Day 8, Day 10, Day 11, and the last day of randomized treatment. For participants who utilized the S/R option, samples were taken on S/R Day 1, S/R Day 3, S/R Day 5, or S/R Day 6, whichever was the last day of S/R treatment. Samples were taken if the participant was symptomatic and continued to be hospitalized on the post-treatment +2, +5, +9, +16 and +28 day assessment. Viral load as measured by PCR. Baseline is defined as the pre-dose value collected on Study Day 1. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: as for outcome 16
Population: IPP Population. Only those participants available at the specified time points were analyzed (represented by n=X, X, X in the category titles)
Measure: Median (Full Range); unit: log10 vp/mL
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 163 | 162 | 163
log10 vp/mL
  Day 3: number analyzed (Participants) | 126 | 127 | 129
  Day 3 | -1.5 [-5.4 to 2.2] | -1.83 [-4.9 to 2.0] | -1.75 [-6.0 to 2.8]
  Day 5: number analyzed (Participants) | 110 | 114 | 114
  Day 5 | -2.51 [-5.8 to 3.2] | -2.71 [-6.2 to 3.1] | -2.73 [-6.3 to 2.3]
  Day 8: number analyzed (Participants) | 15 | 12 | 16
  Day 8 | -2.38 [-4.4 to 1.0] | -3.16 [-5.5 to -0.3] | -1.78 [-5.7 to 1.1]
  Day 10: number analyzed (Participants) | 13 | 6 | 8
  Day 10 | -2.75 [-6.0 to -0.9] | -3.03 [-3.5 to 1.5] | -2.63 [-4.6 to 0.9]
  Day 11: number analyzed (Participants) | 9 | 4 | 7
  Day 11 | -3.58 [-4.9 to -0.6] | -2.6 [-3.1 to 1.7] | -3.29 [-4.9 to -1.0]
  S/R Day 5: number analyzed (Participants) | 0 | 1 | 1
  S/R Day 5 |  | -3.8 [-3.8 to -3.8] | -5.7 [-5.7 to -5.7]
  S/R Day 6: number analyzed (Participants) | 1 | 1 | 2
  S/R Day 6 | -5.2 [-5.2 to -5.2] | -5.4 [-5.4 to -5.4] | -3.84 [-4.0 to -3.7]

18. Secondary Outcome: Number of Participants With no Detectable Viral RNA and the Absence of Cultivable Virus in Lower Respiratory Samples (Bronchoalveolar Lavage Sample [BAL], Endotracheal Aspirate)
Description: Lower respiratory samples included BAL and endotracheal aspirates. Endotracheal aspirates were requested in participants (par.) who were intubated. Upper (nasopharyngeal swabs) and lower (Endotracheal aspirates, bronchoalveolar lavage samples) respiratory samples were collected daily from Baseline/Day 1 through Day 5 and Day 6 (if the last day of randomized treatment [trt]). Endotracheal aspirates were collected in participants who were intubated. If trt was continued beyond Day 5, additional samples were taken on Trt Day 6, Day 8, Day 10, and/or the day of the last dose of randomized trt, if applicable, and S/R Day 1, S/R Day 3, S/R Day 5, or S/R Day 6 if the last day of S/R trt. If the par. was symptomatic and hospitalized, samples were taken on the Post-Trt +2, +5, +9, +16 assessment days, and at the Post-Trt [PT]+28 Day assessment. Assessment of samples was done by quantitative RT-PCR and viral culture.
Time Frame: Baseline (Day 1) and up to 42 days
Population: IPP Population. Data is presented for participants positive at Baseline. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 163 | 162 | 163
Participants
  Influenza A and B Day 1: number analyzed (Participants) | 21 | 17 | 21
  Influenza A and B Day 1 | 0 | 0 | 0
  Influenza A and B Day 2: number analyzed (Participants) | 17 | 15 | 14
  Influenza A and B Day 2 | 0 | 4 | 1
  Influenza A and B Day 3: number analyzed (Participants) | 16 | 10 | 15
  Influenza A and B Day 3 | 1 | 2 | 0
  Influenza A and B Day 4: number analyzed (Participants) | 16 | 10 | 15
  Influenza A and B Day 4 | 2 | 2 | 2
  Influenza A and B Day 5: number analyzed (Participants) | 15 | 10 | 15
  Influenza A and B Day 5 | 3 | 4 | 2
  Influenza A and B Day 6: number analyzed (Participants) | 14 | 5 | 9
  Influenza A and B Day 6 | 3 | 1 | 3
  Influenza A and B Day 8: number analyzed (Participants) | 5 | 3 | 7
  Influenza A and B Day 8 | 2 | 0 | 2
  Influenza A and B Day 10: number analyzed (Participants) | 4 | 3 | 3
  Influenza A and B Day 10 | 0 | 0 | 0
  Influenza A and B S/R Day 1: number analyzed (Participants) | 0 | 0 | 1
  Influenza A and B S/R Day 1 |  |  | 0
  Influenza A and B S/R Day 3: number analyzed (Participants) | 1 | 0 | 1
  Influenza A and B S/R Day 3 | 0 |  | 1
  Influenza A and B S/R Day 5: number analyzed (Participants) | 1 | 0 | 0
  Influenza A and B S/R Day 5 | 0 |  |
  Influenza A and B PT + 2 Days: number analyzed (Participants) | 9 | 3 | 9
  Influenza A and B PT + 2 Days | 4 | 1 | 3
  Influenza A and B PT + 5 Days: number analyzed (Participants) | 11 | 2 | 6
  Influenza A and B PT + 5 Days | 4 | 1 | 0
  Influenza A and B PT + 9 Days: number analyzed (Participants) | 5 | 2 | 4
  Influenza A and B PT + 9 Days | 4 | 1 | 3
  Influenza A and B PT + 16 Days: number analyzed (Participants) | 4 | 1 | 3
  Influenza A and B PT + 16 Days | 3 | 1 | 2
  Influenza A and B PT + 28 Days: number analyzed (Participants) | 1 | 0 | 1
  Influenza A and B PT + 28 Days | 1 |  | 1

19. Secondary Outcome: Median Time to no Detectable Viral RNA and the Absence of Cultivable Virus in Any Obtained Sample (Upper and Lower Respiratory Samples)
Description: Upper (nasopharyngeal swabs) and lower (Endotracheal aspirates, bronchoalveolar lavage samples, where available) respiratory samples were collected daily from Baseline/Day 1 through Day 5 and Day 6 (if the last day of randomized treatment). Endotracheal aspirates were collected in participants who were intubated. If treatment was continued beyond Day 5, additional samples were taken on Treatment Day 6, Day 8, Day 10, and/or the day of the last dose of randomized treatment, if applicable, and S/R Day 1, S/R Day 3, S/R Day 5, or S/R Day 6 if the last day of S/R treatment. If the participant was symptomatic and hospitalized, samples were taken on the Post-treatment+2, +5, +9, +16 assessment days, and at the Post-Treatment +28 Day. Assessment of samples was done by quantitative RT-PCR.
Time Frame: Baseline (Day 1) and up to 42 days
Population: IPP Population. Only those participants available at the specified time points were analyzed. Data also presented for participants positive at Baseline.
Measure: Median (Full Range); unit: Days
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 163 | 162 | 163
Days
  Influenza A and B: number analyzed (Participants) | 114 | 118 | 115
  Influenza A and B | 4 [1 to 34] | 3 [1 to 35] | 4 [1 to 57]
  Positive at Baseline: number analyzed (Participants) | 102 | 104 | 102
  Positive at Baseline | 4 [2 to 34] | 4 [2 to 35] | 4 [2 to 57]

20. Secondary Outcome: Number of Participants With Resistance-associated Mutations Detected in the Neuraminidase (NA) and Hemagglutinin (HA) Gene of Influenza A and B Viruses in Nasopharyngeal Swabs and Endotracheal/BAL Samples
Description: Nasopharyngeal swabs and endotracheal /BAL samples were collected for viral susceptibility analysis. Susceptibility analyses consisted of phenotyping and genotyping. Resistance mutations were detected by genotyping. Viral susceptibility to zanamivir and oral oseltamivir at Baseline and throughout treatment determined by NA and HA (gene of influenza A and B viruses) sequence analysis and NA enzyme inhibition. Number of participants with viral mutation events are summarized, this includes all resistance mutations (substitutions) i.e. those present at Baseline and those that emerged during treatment.
Time Frame: Baseline (Day 1) and up to 42 days
Population: IPP Population
Measure: Count of Participants; unit: Participants
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 163 | 162 | 163
Participants
  NA Gene,H3N2: Y155F | 5 | 7 | 5
  NA Gene,H3N2:S245N | 4 | 4 | 0
  NA Gene,H3N2:I222V | 0 | 1 | 2
  NA Gene,H3N2:N294S/N | 2 | 0 | 0
  NA Gene,H3N2:V149A | 0 | 1 | 1
  NA Gene,H3N2:D198D/G | 0 | 0 | 1
  NA Gene,H3N2:G248G/E | 1 | 0 | 0
  NA Gene,H3N2:N294D/N | 0 | 1 | 0
  NA Gene,H3N2:R292R/K | 0 | 0 | 1
  NA Gene,H3N2:T325I | 1 | 0 | 0
  NA Gene,H3N2:Y155H | 0 | 0 | 1
  NA Gene,H1N1: H275H/Y | 0 | 1 | 4
  NA Gene,H1N1:H275Y | 0 | 1 | 3
  NA Gene,H1N1:Q313R | 1 | 0 | 2
  NA Gene,H1N1:D199N | 1 | 0 | 0
  NA Gene,H1N1:E278G/E | 0 | 0 | 1
  NA Gene,H1N1:I223I/K | 0 | 0 | 1
  NA Gene,H1N1:Q136Q/R | 0 | 0 | 1
  NA Gene,H1N1:S247N | 1 | 0 | 0
  NA Gene,H1N1:S247S/I | 1 | 0 | 0
  NA Gene,H1N1:S247S/N | 0 | 1 | 0
  NA Gene,B: E148G | 1 | 0 | 0
  NA Gene,B: G141E | 0 | 0 | 1
  NA Gene,B: M403I | 1 | 0 | 0
  HA Gene, H3N2:R142G | 18 | 21 | 21
  HA Gene, H3N2:S198A | 13 | 8 | 11
  HA Gene, H3N2:A138S | 3 | 1 | 2
  HA Gene, H3N2:R142K | 0 | 0 | 2
  HA Gene, H3N2:A304A/P | 0 | 0 | 1
  HA Gene, H3N2:A304D | 0 | 1 | 0
  HA Gene, H3N2:L194P/L | 1 | 0 | 0
  HA Gene, H3N2:Q75H | 0 | 1 | 0
  HA Gene, H3N2:S124G | 0 | 0 | 1
  HA Gene, H3N2:S262N | 0 | 1 | 0
  HA Gene, H3N2:H1N1: S183P | 1 | 0 | 2
  HA Gene, H1N1 :D222D/G | 0 | 0 | 2
  HA Gene, H1N1 :D222D/N | 0 | 2 | 0
  HA Gene, H1N1 :D222N | 0 | 0 | 2
  HA Gene, H1N1 :S162N | 0 | 0 | 2
  HA Gene, H1N1 :D187E | 0 | 1 | 0
  HA Gene, H1N1 :D222G | 1 | 0 | 0
  HA Gene, H1N1 :D222S/D/N/G | 1 | 0 | 0
  HA Gene, H1N1 :L151P/L | 0 | 1 | 0
  HA Gene, H1N1 :V152I | 0 | 0 | 1

21. Secondary Outcome: Number of Participants With Any Adverse Event (AE) Considered to be Related to Study Treatment
Description: An AE is defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse, or misuse. All AEs were assessed by the Investigator as related or not related to the study treatment.
Time Frame: Up to 42 days
Population: The Safety Population comprised of all randomized participants who received at least one dose of investigational product and assessed according to their actual treatment received, regardless of the randomization assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 201 | 209 | 205
Participants | 25 | 22 | 35

22. Secondary Outcome: Number of Participants With Any Severe or Grade 3/4 AE
Description: An AE is defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse, or misuse. AEs that occurred during the study were evaluated by the Investigator and graded according to the Division of Acquired Immunodeficiency Syndrome (DAIDS) table for grading the severity of AEs. Grade 3=severe; Grade 4=potentially life threatening.
Time Frame: Up to 42 days
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 201 | 209 | 205
Participants | 39 | 45 | 44

23. Secondary Outcome: Number of Participants Who Permanently Discontinued the Study Treatment Due to an AE
Description: An AE is defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse, or misuse.
Time Frame: Up to 42 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 201 | 209 | 205
Participants | 8 | 10 | 11

24. Secondary Outcome: Number of Participants Who Were Permanently Discontinued From the Study Due to an AE
Description: as for outcome 23
Time Frame: Up to 42 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 201 | 209 | 205
Participants | 14 | 16 | 13

25. Secondary Outcome: Number of Participants With Any Severe or Grade 3/4 Treatment-related AE
Description: An AE is defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse, or misuse. AEs that occurred during the study were evaluated by the Investigator and graded according to the DAIDS table for grading the severity of adult and pediatric AEs. Grade 3=severe; Grade 4=potentially life threatening. All AEs were assessed by the Investigator as related or not related to the study treatment.
Time Frame: Up to 42 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 201 | 209 | 205
Participants | 5 | 3 | 7

26. Secondary Outcome: Number of Participants With the Indicated Chemistry Laboratory Values Shifts From Baseline (Day 1) and up to 42 Days
Description: Samples for laboratory assessments were collected at Baseline (Day 1), Day 3, Day 5/6, Day 8, Day 10/11 (or last day of randomized treatment), switch/rescue (S/R) Day 1, S/R Day 3, and S/R Day 5/6 (last day of S/R treatment for those participants who utilized this option), Post-Treatment +2 (if hospitalized), and Post-Treatment +5, +16, and +28 Days. Clinical chemistry parameters included albumin, alkaline phosphatase (ALP), alanine amino transferase (ALT), aspartate amino tranferase (AST), total bilirubin, calcium, creatine kinase, chloride, carbon dioxide content (CO2), creatinine, potassium, magnesium, sodium. Per the DAIDS table for grading the severity of adult and pediatric AEs, Grade (G) 1=mild, G2= moderate, G3=severe and G4=potentially life threatening. The number of participants with values that were G1, G2, G3 and G4 relative to the normal range are summarized.
Time Frame: Baseline (Day 1) and up to 42 days
Population: Safety Population. Only the participants available at the time of assessment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 201 | 209 | 205
Participants
  Albumin G1: number analyzed (Participants) | 194 | 203 | 202
  Albumin G1 | 12 | 18 | 15
  Albumin G2: number analyzed (Participants) | 194 | 203 | 202
  Albumin G2 | 32 | 43 | 40
  Albumin G3: number analyzed (Participants) | 194 | 203 | 202
  Albumin G3 | 1 | 5 | 0
  Albumin G4: number analyzed (Participants) | 194 | 203 | 202
  Albumin G4 | 0 | 0 | 0
  ALP G1: number analyzed (Participants) | 194 | 203 | 202
  ALP G1 | 10 | 15 | 9
  ALP G2: number analyzed (Participants) | 194 | 203 | 202
  ALP G2 | 0 | 4 | 1
  ALP G3: number analyzed (Participants) | 194 | 203 | 202
  ALP G3 | 0 | 2 | 0
  ALP G4: number analyzed (Participants) | 194 | 203 | 202
  ALP G4 | 0 | 0 | 0
  ALT G1: number analyzed (Participants) | 194 | 203 | 202
  ALT G1 | 13 | 10 | 12
  ALT G2: number analyzed (Participants) | 194 | 203 | 202
  ALT G2 | 2 | 1 | 1
  ALT G3: number analyzed (Participants) | 194 | 203 | 202
  ALT G3 | 0 | 0 | 0
  ALT G4: number analyzed (Participants) | 194 | 203 | 202
  ALT G4 | 0 | 0 | 1
  AST G1: number analyzed (Participants) | 193 | 202 | 202
  AST G1 | 23 | 27 | 19
  AST G2: number analyzed (Participants) | 193 | 202 | 202
  AST G2 | 8 | 8 | 6
  AST G3: number analyzed (Participants) | 193 | 202 | 202
  AST G3 | 2 | 0 | 2
  AST G4: number analyzed (Participants) | 193 | 202 | 202
  AST G4 | 0 | 0 | 1
  Total Bilirubin G1: number analyzed (Participants) | 194 | 203 | 202
  Total Bilirubin G1 | 5 | 2 | 2
  Total Bilirubin G2: number analyzed (Participants) | 194 | 203 | 202
  Total Bilirubin G2 | 3 | 2 | 3
  Total Bilirubin G3: number analyzed (Participants) | 194 | 203 | 202
  Total Bilirubin G3 | 1 | 2 | 0
  Total Bilirubin G4: number analyzed (Participants) | 194 | 203 | 202
  Total Bilirubin G4 | 0 | 0 | 1
  Creatine Kinase G1: number analyzed (Participants) | 194 | 203 | 202
  Creatine Kinase G1 | 10 | 11 | 6
  Creatine Kinase G2: number analyzed (Participants) | 194 | 203 | 202
  Creatine Kinase G2 | 3 | 3 | 6
  Creatine Kinase G3: number analyzed (Participants) | 194 | 203 | 202
  Creatine Kinase G3 | 1 | 2 | 4
  Creatine Kinase G4: number analyzed (Participants) | 194 | 203 | 202
  Creatine Kinase G4 | 1 | 1 | 2
  CO2 G1: number analyzed (Participants) | 193 | 202 | 202
  CO2 G1 | 34 | 43 | 47
  CO2 G2,: number analyzed (Participants) | 193 | 202 | 202
  CO2 G2, | 4 | 9 | 6
  CO2 G3: number analyzed (Participants) | 193 | 202 | 202
  CO2 G3 | 0 | 0 | 0
  CO2 G4: number analyzed (Participants) | 193 | 202 | 202
  CO2 G4 | 0 | 1 | 0
  Creatinine G1: number analyzed (Participants) | 194 | 203 | 202
  Creatinine G1 | 6 | 5 | 4
  Creatinine G2: number analyzed (Participants) | 194 | 203 | 202
  Creatinine G2 | 11 | 7 | 4
  Creatinine G3: number analyzed (Participants) | 194 | 203 | 202
  Creatinine G3 | 8 | 7 | 4
  Creatinine G4: number analyzed (Participants) | 194 | 203 | 202
  Creatinine G4 | 0 | 0 | 1
  Magnesium G1: number analyzed (Participants) | 194 | 203 | 202
  Magnesium G1 | 14 | 14 | 15
  Magnesium G2,: number analyzed (Participants) | 194 | 203 | 202
  Magnesium G2, | 7 | 9 | 4
  Magnesium G3: number analyzed (Participants) | 194 | 203 | 202
  Magnesium G3 | 0 | 0 | 0
  Magnesium G4: number analyzed (Participants) | 194 | 203 | 202
  Magnesium G4 | 0 | 0 | 0
  Hypercalcemia G1: number analyzed (Participants) | 193 | 202 | 202
  Hypercalcemia G1 | 0 | 0 | 0
  Hypercalcemia G2: number analyzed (Participants) | 193 | 202 | 202
  Hypercalcemia G2 | 0 | 0 | 0
  Hypercalcemia G3: number analyzed (Participants) | 193 | 202 | 202
  Hypercalcemia G3 | 0 | 0 | 0
  Hypercalcemia G4: number analyzed (Participants) | 193 | 202 | 202
  Hypercalcemia G4 | 0 | 0 | 0
  Hyperkalemia G1: number analyzed (Participants) | 193 | 202 | 202
  Hyperkalemia G1 | 0 | 1 | 1
  Hyperkalemia G2: number analyzed (Participants) | 193 | 202 | 202
  Hyperkalemia G2 | 0 | 0 | 0
  Hyperkalemia G3: number analyzed (Participants) | 193 | 202 | 202
  Hyperkalemia G3 | 0 | 0 | 0
  Hyperkalemia G4: number analyzed (Participants) | 193 | 202 | 202
  Hyperkalemia G4 | 1 | 0 | 1
  Hypernatremia G1: number analyzed (Participants) | 194 | 203 | 202
  Hypernatremia G1 | 4 | 10 | 4
  Hypernatremia G2: number analyzed (Participants) | 194 | 203 | 202
  Hypernatremia G2 | 1 | 1 | 0
  Hypernatremia G3: number analyzed (Participants) | 194 | 203 | 202
  Hypernatremia G3 | 0 | 1 | 1
  Hypernatremia G4: number analyzed (Participants) | 194 | 203 | 202
  Hypernatremia G4 | 0 | 0 | 0
  Hypocalcemia G1: number analyzed (Participants) | 193 | 202 | 202
  Hypocalcemia G1 | 43 | 48 | 40
  Hypocalcemia G2: number analyzed (Participants) | 193 | 202 | 202
  Hypocalcemia G2 | 26 | 39 | 42
  Hypocalcemia G3: number analyzed (Participants) | 193 | 202 | 202
  Hypocalcemia G3 | 7 | 8 | 8
  Hypocalcemia G4: number analyzed (Participants) | 193 | 202 | 202
  Hypocalcemia G4 | 0 | 1 | 0
  Hypokalemia G1: number analyzed (Participants) | 193 | 202 | 202
  Hypokalemia G1 | 16 | 12 | 21
  Hypokalemia G2: number analyzed (Participants) | 193 | 202 | 202
  Hypokalemia G2 | 1 | 1 | 1
  Hypokalemia G3: number analyzed (Participants) | 193 | 202 | 202
  Hypokalemia G3 | 1 | 0 | 0
  Hypokalemia G4: number analyzed (Participants) | 193 | 202 | 202
  Hypokalemia G4 | 0 | 0 | 0
  Hyponatremia G1: number analyzed (Participants) | 194 | 203 | 202
  Hyponatremia G1 | 42 | 34 | 26
  Hyponatremia G2: number analyzed (Participants) | 194 | 203 | 202
  Hyponatremia G2 | 2 | 2 | 4
  Hyponatremia G3: number analyzed (Participants) | 194 | 203 | 202
  Hyponatremia G3 | 0 | 2 | 0
  Hyponatremia G4: number analyzed (Participants) | 194 | 203 | 202
  Hyponatremia G4 | 0 | 0 | 1

27. Secondary Outcome: Number of Participants With the Indicated Hematology Values Shifts From Baseline (Day 1) and up to 42 Days
Description: Blood samples for laboratory assessments were collected at Baseline (Day 1), Day 3, Day 5/6, Day 8, Day 10/11 (or last day of randomized treatment), S/R Day 1, S/R Day 3, and S/R Day 5/6 (last day of S/R treatment for those participants who utilized this option), Post-Treatment +2 (if hospitalized), and Post-Treatment +5, +16, and +28 Days. Hematology parameters included hemoglobin, lymphocytes, total neutrophils, platelet count, and white blood cell (WBC) count. Per the DAIDS table for grading the severity of adult and pediatric AEs, Grade (G) 1=mild, G2= moderate, G3=severe and G4=potentially life threatening. The number of participants with values that were G1, G2, G3 and G4 relative to the normal range for the indicated hematology parameters is summarized. Baseline is defined as the pre-dose value collected on Study Day 1.
Time Frame: Baseline (Day 1) and up to 42 days
Population: Safety Population. Only the participants available at the time of assessment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 201 | 209 | 205
Participants
  Hemoglobin G1: number analyzed (Participants) | 194 | 202 | 200
  Hemoglobin G1 | 28 | 25 | 28
  Hemoglobin G2: number analyzed (Participants) | 194 | 202 | 200
  Hemoglobin G2 | 11 | 19 | 13
  Hemoglobin G3: number analyzed (Participants) | 194 | 202 | 200
  Hemoglobin G3 | 14 | 10 | 8
  Hemoglobin G4: number analyzed (Participants) | 194 | 202 | 200
  Hemoglobin G4 | 0 | 4 | 1
  Lymphocytes G1: number analyzed (Participants) | 186 | 199 | 198
  Lymphocytes G1 | 8 | 18 | 10
  Lymphocytes G2: number analyzed (Participants) | 186 | 199 | 198
  Lymphocytes G2 | 11 | 15 | 11
  Lymphocytes G3: number analyzed (Participants) | 186 | 199 | 198
  Lymphocytes G3 | 16 | 21 | 18
  Lymphocytes G4: number analyzed (Participants) | 186 | 199 | 198
  Lymphocytes G4 | 18 | 19 | 14
  Neutrophils G1: number analyzed (Participants) | 193 | 202 | 200
  Neutrophils G1 | 2 | 2 | 3
  Neutrophils G2: number analyzed (Participants) | 193 | 202 | 200
  Neutrophils G2 | 2 | 0 | 0
  Neutrophils G3: number analyzed (Participants) | 193 | 202 | 200
  Neutrophils G3 | 0 | 1 | 0
  Neutrophils G4: number analyzed (Participants) | 193 | 202 | 200
  Neutrophils G4 | 1 | 0 | 3
  Platelets G1: number analyzed (Participants) | 194 | 200 | 198
  Platelets G1 | 8 | 22 | 21
  Platelets G2: number analyzed (Participants) | 194 | 200 | 198
  Platelets G2 | 18 | 12 | 16
  Platelets G3: number analyzed (Participants) | 194 | 200 | 198
  Platelets G3 | 4 | 3 | 2
  Platelets G4: number analyzed (Participants) | 194 | 200 | 198
  Platelets G4 | 2 | 1 | 2
  Leukocytes G1: number analyzed (Participants) | 194 | 202 | 200
  Leukocytes G1 | 3 | 2 | 1
  Leukocytes G2: number analyzed (Participants) | 194 | 202 | 200
  Leukocytes G2 | 3 | 5 | 3
  Leukocytes G3: number analyzed (Participants) | 194 | 202 | 200
  Leukocytes G3 | 0 | 1 | 0
  Leukocytes G4: number analyzed (Participants) | 194 | 202 | 200
  Leukocytes G4 | 1 | 0 | 2

28. Secondary Outcome: Number of Participants With the Indicated Treatment-emergent (TE) Grade (G) 3/4 Clinical Chemistry Toxicities
Description: A toxicity was considered to be TE if it was greater than the Baseline grade, and if it had developed or increased post-Baseline in intensity (and prior to the last dose of investigational product). Clinical chemistry parameters included albumin, ALP, ALT, AST, total bilirubin, calcium, creatine kinase, chloride, CO2/bicarbonate, creatinine, potassium, magnesium and sodium. Per the DAIDS table for grading the severity of adult and pediatric AEs, Grade 3=severe and Grade 4=potentially life threatening. Baseline is defined as the pre-dose value collected on Study Day 1.
Time Frame: Baseline (Day 1) and up to 42 days
Population: Safety population. Only the participants available at the time of assessment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 201 | 209 | 205
Participants
  Albumin, G3: number analyzed (Participants) | 194 | 203 | 202
  Albumin, G3 | 6 | 3 | 4
  Albumin, G4: number analyzed (Participants) | 194 | 203 | 202
  Albumin, G4 | 0 | 0 | 0
  ALP, G3: number analyzed (Participants) | 194 | 203 | 202
  ALP, G3 | 0 | 2 | 0
  ALP, G4: number analyzed (Participants) | 194 | 203 | 202
  ALP, G4 | 1 | 0 | 1
  ALT, G3: number analyzed (Participants) | 194 | 203 | 202
  ALT, G3 | 2 | 2 | 4
  ALT, G4: number analyzed (Participants) | 194 | 203 | 202
  ALT, G4 | 0 | 2 | 1
  AST, G3: number analyzed (Participants) | 193 | 202 | 202
  AST, G3 | 2 | 4 | 5
  AST, G4: number analyzed (Participants) | 193 | 202 | 202
  AST, G4 | 1 | 2 | 1
  Total Bilirubin, G3: number analyzed (Participants) | 194 | 203 | 202
  Total Bilirubin, G3 | 2 | 2 | 1
  Total Bilirubin, G4: number analyzed (Participants) | 194 | 203 | 202
  Total Bilirubin, G4 | 0 | 0 | 0
  Creatine Kinase, G3 | 2 | 3 | 2
  Creatine Kinase, G4: number analyzed (Participants) | 194 | 203 | 202
  Creatine Kinase, G4 | 3 | 1 | 1
  Carbon Dioxide, G3: number analyzed (Participants) | 193 | 202 | 202
  Carbon Dioxide, G3 | 0 | 0 | 0
  Carbon Dioxide, G4: number analyzed (Participants) | 193 | 202 | 202
  Carbon Dioxide, G4 | 1 | 0 | 0
  Creatinine, G3: number analyzed (Participants) | 194 | 203 | 202
  Creatinine, G3 | 3 | 6 | 1
  Creatinine, G4: number analyzed (Participants) | 194 | 203 | 202
  Creatinine, G4 | 3 | 2 | 0
  Magnesium, G3: number analyzed (Participants) | 194 | 203 | 202
  Magnesium, G3 | 1 | 0 | 0
  Magnesium, G4: number analyzed (Participants) | 194 | 203 | 202
  Magnesium, G4 | 0 | 0 | 1
  Hypercalcemia, G3: number analyzed (Participants) | 194 | 202 | 202
  Hypercalcemia, G3 | 0 | 0 | 0
  Hypercalcemia, G4: number analyzed (Participants) | 194 | 202 | 202
  Hypercalcemia, G4 | 0 | 0 | 0
  Hyperkalemia, G3: number analyzed (Participants) | 193 | 202 | 202
  Hyperkalemia, G3 | 2 | 0 | 1
  Hyperkalemia, G4: number analyzed (Participants) | 193 | 202 | 202
  Hyperkalemia, G4 | 1 | 5 | 3
  Hypernatremia, G3: number analyzed (Participants) | 194 | 203 | 202
  Hypernatremia, G3 | 0 | 1 | 5
  Hypernatremia, G4: number analyzed (Participants) | 194 | 203 | 202
  Hypernatremia, G4 | 0 | 0 | 0
  Hypocalcemia, G3: number analyzed (Participants) | 193 | 202 | 202
  Hypocalcemia, G3 | 10 | 7 | 8
  Hypocalcemia, G4: number analyzed (Participants) | 193 | 202 | 202
  Hypocalcemia, G4 | 2 | 4 | 4
  Hypokalemia, G3: number analyzed (Participants) | 193 | 202 | 202
  Hypokalemia, G3 | 0 | 0 | 0
  Hypokalemia, G4: number analyzed (Participants) | 193 | 202 | 202
  Hypokalemia, G4 | 0 | 0 | 0
  Hyponatremia, G3: number analyzed (Participants) | 194 | 203 | 202
  Hyponatremia, G3 | 1 | 0 | 0
  Hyponatremia G4: number analyzed (Participants) | 194 | 203 | 202
  Hyponatremia G4 | 0 | 0 | 0

29. Secondary Outcome: Number of Participants With the Indicated Treatment-emergent (TE) Grade 3/4 Hematology Toxicities
Description: A toxicity was considered to be TE if it was greater than the Baseline grade, and if it had developed or increased post-Baseline in intensity (and prior to the last dose of investigational product). The hematology parameters included hemoglobin, lymphocytes, total neutrophils, platelet count, and WBC count. Per the DAIDS table for grading the severity of adult and pediatric AEs, Grade 3=severe and Grade 4=potentially life threatening. Baseline is defined as the pre-dose value collected on Study Day 1.
Time Frame: Baseline (Day 1) and up to 42 days
Population: Safety Population. Only the participants available at the time of assessment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 201 | 209 | 205
Participants
  Hemoglobin, G3: number analyzed (Participants) | 194 | 202 | 200
  Hemoglobin, G3 | 29 | 24 | 26
  Hemoglobin, G4: number analyzed (Participants) | 194 | 202 | 200
  Hemoglobin, G4 | 2 | 5 | 8
  Lymphocytes, G3: number analyzed (Participants) | 186 | 199 | 198
  Lymphocytes, G3 | 6 | 5 | 11
  Lymphocytes, G4: number analyzed (Participants) | 186 | 199 | 198
  Lymphocytes, G4 | 3 | 14 | 7
  Total Neutrophils, G3: number analyzed (Participants) | 193 | 202 | 200
  Total Neutrophils, G3 | 1 | 2 | 2
  Total Neutrophils, G4: number analyzed (Participants) | 193 | 202 | 200
  Total Neutrophils, G4 | 4 | 4 | 3
  Platelet count, G3: number analyzed (Participants) | 194 | 200 | 198
  Platelet count, G3 | 4 | 4 | 5
  Platelet count, G4: number analyzed (Participants) | 194 | 200 | 198
  Platelet count, G4 | 3 | 3 | 2
  Leukocytes Count, G3: number analyzed (Participants) | 194 | 202 | 200
  Leukocytes Count, G3 | 1 | 1 | 0
  Leukocytes Count, G4: number analyzed (Participants) | 194 | 202 | 200
  Leukocytes Count, G4 | 2 | 1 | 3

30. Secondary Outcome: Median Quantity of Oxygen Delivery Measured at Baseline (Day 1) and During the Study
Description: Oxygen delivery were assessed three times daily at Baseline (Day 1) and during the treatment period/hospitalization (ideally at least 6 hours apart) and once daily during inpatient/hospitalization and once at Post +5 days, +16 days, and +28 days clinic visits. The median quantity of oxygen delivery during the study was not summarized since the data was not collected in a way to accurately calculate values. Baseline is defined as the pre-dose value collected on Study Day 1.
Time Frame: Baseline (Day 1) and during the study
Population: This end point was not analyzed
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 0 | 0 | 0

31. Secondary Outcome: Number of Participants Assessed as Normal/Abnormal (Clinically Significant [CS] and Not Clinically Significant [NCS]) for 12-lead Electrocardiogram (ECG) at Baseline (Day 1) and Day 4
Description: On Baseline/Day 1, a 12-lead ECG was obtained within approximately 24 hours prior to dosing. The number of participants with an ECG status of normal and abnormal CS or NCS, as determined by the Investigator, is reported. Normal=all ECG parameters within the accepted normal ranges. Abnormal=ECG findings outside of normal ranges. CS=ECG with a CS abnormality that meets exclusion criteria. NCS=ECG with an abnormality that is not CS nor meets exclusion criteria, per Investigator, based on reasonable standards of clinical judgment. In the original protocol ECGs were also done on Day 4, however, amendment 2 removed this requirement and therefore not all participants had Day 4 ECGs.
Time Frame: Baseline (Day 1) and Day 4
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 197 | 208 | 203
Participants
  Normal | 100 | 121 | 99
  Abnormal - Not Clinically Significant | 97 | 86 | 102
  Abnormal - Clinically Significant | 5 | 4 | 7

32. Secondary Outcome: Serum Concentration of IV Zanamivir
Description: Pharmacokinetic samples were collected at four time points to characterize peak concentration (end of infusion; C[EOI]) after the first dose on Day 1 and on Day 4 to characterize the pre-dose concentration (C[0]), the peak concentration C(EOI), and the trough concentration at 11-12 hours post-dose (C[12]) of zanamavir. Data was summarized by Creatinine clearance (CL) Category. The dose on Day 1 is the initial dose (unadjusted) and the dose on Day 4 is the maintenance dose.
Time Frame: Day 1 and Day 4
Population: Pharmacokinetic (PK) Population comprised of all participants who received IV zanamivir and underwent sparse PK sampling during the study from which one or more serum zanamivir concentrations was determined. This outcome was not analyzed for participants receiving oseltamivir 75 mg. Only the participants available at the time point were analyzed.
Measure: Mean (Standard Deviation); unit: microgram/Liter (mcg/L)
Arm/Group | IV Zanamivir 300 mg | IV Zanamivir 600 mg | Oral Oseltamivir 75 mg
Number analyzed (Participants) | 180 | 187 | 0
microgram/Liter (mcg/L)
  CL <15, Day 1, 30 min: number analyzed (Participants) | 1 | 3 | 0
  CL <15, Day 1, 30 min | 14454.6 (NA) — Data not collected | 26410.8 (21335.43) |
  CL <15, Day 4, pre-dose: number analyzed (Participants) | 1 | 2 | 0
  CL <15, Day 4, pre-dose | 293.2 (NA) — Data not collected | 9635.6 (8270.67) |
  CL <15, Day 4, 30 min: number analyzed (Participants) | 1 | 1 | 0
  CL <15, Day 4, 30 min | 1329.4 (NA) — Data not collected | 19828.9 (NA) — Data not available |
  CL <15, Day 4, 11-12 hr: number analyzed (Participants) | 1 | 1 | 0
  CL <15, Day 4, 11-12 hr | 605.1 (NA) — Data not collected | 15459.1 (NA) — Data not available |
  CL 15-<30, Day 13, 30 min: number analyzed (Participants) | 13 | 9 | 0
  CL 15-<30, Day 13, 30 min | 20403.3 (11623.28) | 41102.8 (13884.08) |
  CL 15-<30, Day 4, pre-dose: number analyzed (Participants) | 10 | 6 | 0
  CL 15-<30, Day 4, pre-dose | 5906.4 (7167.87) | 4995.6 (1966.72) |
  CL 15-<30, Day 4, 30 min: number analyzed (Participants) | 10 | 6 | 0
  CL 15-<30, Day 4, 30 min | 13636.4 (14029.44) | 13378 (2581.36) |
  CL 15-<30, Day 4, 11-12 hr: number analyzed (Participants) | 8 | 5 | 0
  CL 15-<30, Day 4, 11-12 hr | 7600.3 (8061.65) | 4953.4 (2232.16) |
  CL 30-<50, Day 1, 30 min: number analyzed (Participants) | 28 | 18 | 0
  CL 30-<50, Day 1, 30 min | 18756.8 (12806.43) | 42467.3 (14574.82) |
  CL 30-<50, Day 4, pre-dose: number analyzed (Participants) | 12 | 15 | 0
  CL 30-<50, Day 4, pre-dose | 2094.8 (1300.99) | 7637.4 (7212.1) |
  CL 30-<50, Day 4, 30 min: number analyzed (Participants) | 12 | 13 | 0
  CL 30-<50, Day 4, 30 min | 12334.4 (12121.18) | 159292.1 (473267.3) |
  CL 30-<50, Day 4, 11-12 hr: number analyzed (Participants) | 11 | 13 | 0
  CL 30-<50, Day 4, 11-12 hr | 2932.5 (2425.81) | 19549.2 (40577.76) |
  CL 50-<80, Day 1, 30 min: number analyzed (Participants) | 36 | 49 | 0
  CL 50-<80, Day 1, 30 min | 19146.7 (8853.11) | 49666.1 (111785.9) |
  CL 50-<80, Day 4, pre-dose: number analyzed (Participants) | 31 | 25 | 0
  CL 50-<80, Day 4, pre-dose | 2793.3 (4694.43) | 13107.7 (33768.61) |
  CL 50-<80, Day 4, 30 min: number analyzed (Participants) | 32 | 25 | 0
  CL 50-<80, Day 4, 30 min | 31541.3 (93381) | 22220.4 (10064.83) |
  CL 50-<80, Day 4, 11-12 hr: number analyzed (Participants) | 30 | 23 | 0
  CL 50-<80, Day 4, 11-12 hr | 1345.9 (1122.18) | 22623.9 (57663.24) |
  CL >=80, Day 1, 30 min,: number analyzed (Participants) | 93 | 96 | 0
  CL >=80, Day 1, 30 min, | 18561.7 (10332.14) | 35139.2 (17693.85) |
  CL >=80, Day 4, pre-dose: number analyzed (Participants) | 99 | 107 | 0
  CL >=80, Day 4, pre-dose | 2342.6 (6672.12) | 19379.8 (105056.3) |
  CL >=80, Day 4, 30 min: number analyzed (Participants) | 100 | 106 | 0
  CL >=80, Day 4, 30 min | 21580.7 (22062.69) | 75255.1 (167670.6) |
  CL >=80, Day 4, 11-12 hr: number analyzed (Participants) | 94 | 99 | 0
  CL >=80, Day 4, 11-12 hr | 2036.2 (4412.75) | 19428.7 (142284.7) |
  Missing, Day 1, 30 min: number analyzed (Participants) | 0 | 2 | 0
  Missing, Day 1, 30 min |  | 41109.7 (3831.74) |

ADVERSE EVENTS:
Time Frame: From the start of study drug until follow-up (up to 42 days).
Description: Safety population was used to assess adverse events.
Arm/Group | Intravenous (IV) Zanamivir 300mg Twice Daily | Intravenous (IV) Zanamivir 600mg Twice Daily | Oral Oseltamivir 75mg Twice Daily
All-Cause Mortality (participants affected / at risk) | 15/201 | 15/209 | 11/205
Serious Adverse Events (participants affected / at risk) | 38/201 | 33/209 | 38/205
Other Adverse Events (participants affected / at risk) | 17/201 | 26/209 | 24/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous (IV) Zanamivir 300mg Twice Daily (N=201) | Intravenous (IV) Zanamivir 600mg Twice Daily (N=209) | Oral Oseltamivir 75mg Twice Daily (N=205)
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Distributive shock (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 0
Mechanical ventilation (Surgical and medical procedures) | 1 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Anti-neutrophil cytoplasmic antibody (Immune system disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 2 | 2 | 2
Catheter site haemorrhage (General disorders) | 1 | 0 | 0
Hyperthermia (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Delirium febrile (Psychiatric disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
ECG signs of ventricular hypertrophy (Investigations) | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1
Hypoalbuminaemia (Investigations) | 1 | 0 | 0
Hypocalcaemia (Investigations) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 2 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 5
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0
Chronic obstructive pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory disorderv (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Disseminated intravascular (Blood and lymphatic system disorders) | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Neuromyopathy (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0
IgA nephropathy (Renal and urinary disorders) | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 7 | 1 | 4
Septic shock (Infections and infestations) | 4 | 1 | 2
Sepsis (Infections and infestations) | 1 | 1 | 1
Bronchitis (Infections and infestations) | 2 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 1
Pneumonia necrotising (Infections and infestations) | 0 | 1 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous (IV) Zanamivir 300mg Twice Daily (N=201) | Intravenous (IV) Zanamivir 600mg Twice Daily (N=209) | Oral Oseltamivir 75mg Twice Daily (N=205)
Diarrhoea (Gastrointestinal disorders) | 10 | 15 | 14
Constipation (Gastrointestinal disorders) | 7 | 13 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.